CLINICAL TRIAL: NCT06167200
Title: Validation of a Clinical Complications Scale (CCS) in Patients With Disorders of Consciousness
Acronym: SCC_DOC
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Anna Estraneo, Neurologist, Senior Researcher, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: SCC_DOC
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Disorders of Consciousness
Keywords: Disorders of Consciousness; clinical complications
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with DoC consecutively admitted to participating units and met the inclusion criteria: Patients in VS or MCS due to severe acquired brain injury with different etiology (traumatic, anoxic, vascular) consecutively admitted at participating neurorehabilitation units. The total sample will be composed of 42 patients (n=7 pts per participating unit).
  Interventions: Other: No intervention, study is observational

INTERVENTIONS:
Other: No intervention, study is observational — No intervention, study is observational

SUMMARY:
The clinical condition of severe cognitive-motor impairment of Disorders of Consciousness (DoC; e.g., Vegetative State - VS, and Minimal Consciousness State - MCS), is characterized by a high risk of developing clinical complications. In this study, the investigators propose a new Clinical Complications Scale (CCS) developed to assess the impact of clinical complications on the long-term evolution of a cohort of patients with DoC.

This is a multi-site prospective observational study conducted in patients with Severe Acquired Brain Injury and DoC admitted to six centers of Fondazione Don Gnocchi (Italy), with clinical data collection not deviating from routine practice (except for CCS administration). The study is non-commercial and will have a maximum total duration of 24 months. It is planned to assess inter-rater agreement and concurrent validity with a similar instrument (CoCoS scale).

DETAILED DESCRIPTION:
Validation of a scale for the assessment of clinical complications (Clinical Complications Scale, CCS) on a sample of DoC patients with:

* assessment of inter-rater agreement;
* assessment of concurrent validity with a similar instrument (CoCoS).

This study will be implemented throutgh three phases:

(i) Identification of a group of evaluators at participating centers (n=3 per center; total n=18) and training them to administer the CCS and CoCos scales by group videoconference; (ii) Recruitment of a sample of DoC patients (n=7 per center; total n=42) who will each undergo assessment with CCS (administered twice by two independent assessors, A and B) and with CoCoS (administered by a third independent assessor, C); (iii) Evaluation of the degree of agreement between observers in administering the CCS scale (agreement between evaluators A and B) and evaluation of concurrent validity between CCS and CoCoS scale (agreement between evaluators A/B and C).

The study involves the collection of the following clinical data for each patient on admission and during the following 15 days:

* Demographic data respecting patient anonymity (patient's numeric identification code, age, sex, ethnicity, education);
* Anamnestic data (date and etiology of acute event);
* Clinical data including blood chemistry tests, clinical complications and related therapies administered as per normal clinical reports in use at enrolling units, and referring to the 15-day period following the date of enrollment. Each patient also will be evaluated with CRS-R scale 3-5 times within one week after enrollment for confirmation of the diagnosis of DoC. Assessments with CCS and CoCoS clinical scales completed on clinical reports referring to medical complications that occurred within 15 days of enrollment.

The CCS provides a record of clinical complications in 11 categories corresponding to systems of the body (metabolic abnormalities, disorders-cardiovascular, skin and musculoskeletal problems, gastrointestinal disorders, genito-urinary disorders, respiratory disorders) or categories of clinical problems frequently encountered in the population of patients with DoC (neurosurgical complications, epilepsy and myoclonus, paraosteortropathy, neurovegetative crisis, sepsis; Estraneo et al., 2018). For each category, the severity of complications is graded from 0 (absent complication) to 3 (severe complication) based on the intensity of the therapeutic intervention required, interference with the clinic, and/or frequency and duration of morbid events (an exception is the "sepsis" category for which only presence/absence is recorded). In the case of multiple clinical complications occurring within the same category, the most severe will be considered for the severity score. In this way, a cumulative scale score with range 0-31 can be derived.

Descriptive data from the sample at study entry will be expressed in terms of mean and standard deviation for quantitative variables and as frequencies for nominal variables. For the assessment of inter-rater agreement in the administration of the CCS, Fleiss' weighted K-index will be calculated on the individual subscale scores and the total score of the scale administered to each patient by two different operators. For concurrent validity testing between the CCS and CoCoS scales, Fleiss' weighted K-index will be calculated between the scores at the subscales in common between the two instruments, while Spearman's correlation coefficient for ranks will be calculated on the total scores obtained by patients on the two scales.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of VS or MCS, in accordance with international standard diagnostic criteria (Giacino et al., 2002) and confirmed by Coma Recovery Scale-Revised (CRS-R; Giacino et al., 2004) assessment repeated 3-5 times within a week (Wannez et al., 2017);
* Time post-injury ≥28 days;
* age ≥18 years;
* Traumatic, vascular, anoxic, or mixed etiology.

Exclusion Criteria:

* Absence of the informed consent by the patient's legal representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in VS or MCS due to severe acquired brain injury with different etiology (traumatic, anoxic, vascular) consecutively admitted at participating neurorehabilitation units. The total sample will be composed of 42 patients (n=7 pts per participating unit).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
inter-rater reliability | 15 days from enrolment
  agreement in scores between different examiners
concurrent validity | 15 days from enrolment
  correlation between scores on the CCS and the CoCoS

CONTACTS AND LOCATIONS:
Overall Officials: Anna Estraneo, MD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (6):
- Italy (6):
  - Polo Specialistico Riabilitativo Fondazione Don Carlo Gnocchi ONLUS, Sant'Angelo dei Lombardi, Avellino
  - IRCCS Fondazione Don Carlo Gnocchi Firenze, Florence
  - Polo Riabilitativo del Levante Ligure Fondazione Don Gnocchi, La Spezia
  - IRCCS S. Maria Nascente Fondazione Don Gnocchi, Milan
  - Istituto Palazzolo Fondazione Don Gnocchi, Milan
  - Centro Spalenza Fondazione Don Gnocchi, Rovato

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giacino JT, Ashwal S, Childs N, Cranford R, Jennett B, Katz DI, Kelly JP, Rosenberg JH, Whyte J, Zafonte RD, Zasler ND. The minimally conscious state: definition and diagnostic criteria. Neurology. 2002 Feb 12;58(3):349-53. doi: 10.1212/wnl.58.3.349. PMID 11839831
- [Background] Wannez S, Heine L, Thonnard M, Gosseries O, Laureys S; Coma Science Group collaborators. The repetition of behavioral assessments in diagnosis of disorders of consciousness. Ann Neurol. 2017 Jun;81(6):883-889. doi: 10.1002/ana.24962. PMID 28543735
- [Background] Pistoia F, Carolei A, Bodien YG, Greenfield S, Kaplan S, Sacco S, Pistarini C, Casalena A, De Tanti A, Cazzulani B, Bellaviti G, Sara M, Giacino J. The Comorbidities Coma Scale (CoCoS): Psychometric Properties and Clinical Usefulness in Patients With Disorders of Consciousness. Front Neurol. 2019 Oct 17;10:1042. doi: 10.3389/fneur.2019.01042. eCollection 2019. PMID 31681139
- [Background] Estraneo A, Loreto V, Masotta O, Pascarella A, Trojano L. Do Medical Complications Impact Long-Term Outcomes in Prolonged Disorders of Consciousness? Arch Phys Med Rehabil. 2018 Dec;99(12):2523-2531.e3. doi: 10.1016/j.apmr.2018.04.024. Epub 2018 May 26. PMID 29807003
- [Background] Giacino JT, Kalmar K, Whyte J. The JFK Coma Recovery Scale-Revised: measurement characteristics and diagnostic utility. Arch Phys Med Rehabil. 2004 Dec;85(12):2020-9. doi: 10.1016/j.apmr.2004.02.033. PMID 15605342